CLINICAL TRIAL: NCT05618132
Title: Stepwise Treatment and Acetylcholine Rechallenge in Vasospastic Angina to Guide Patient-tailored Treatment
Brief Title: ReACHallenge Trial: Acetylcholine Rechallenge After Pretreatment With Vasoactive Drugs
Acronym: ReACHallenge
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2806
Record Dates: First submitted 2022-11-08; First posted 2022-11-16 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2022-10

CONDITIONS: Angina Pectoris, Variant; Angina Pectoris; Spasm-Induced; Angina Pectoris With Normal Coronary Arteriogram
Keywords: Vasospastic angina; Angina with non-obstructive coronary arteries (ANOCA); Acetylcholine
MeSH Terms: conditions — Angina Pectoris, Variant; Angina Pectoris; Microvascular Angina

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vasospastic angina (Experimental): Interventional diagnostic protocol
  Interventions: Diagnostic Test: Acetylcholine rechallenge

INTERVENTIONS:
Diagnostic Test: Acetylcholine rechallenge — STEP 1 consists of verapamil 1mg IC. Angiography after 60 seconds, if spasm persists, NTG 200µg IC is given (step 2). If verapamil suppresses spasm, ACH rechallenge (ACHR) is performed after 3 minutes.
  In STEP 2, patients with persistent spasm after verapamil or with spasm after ACHR receive NTG 200µg IC. Angiography after 60 seconds, if spasm persists, NTG 200µg IC is delivered again. If refractory spasm occurs, atropine 1mg IV is given. Coronary spasm is considered suppressed once ACHR can no longer provoke spasm. NTG 200µg IC is given as final drug regardless of spasm.
  ACHR consists of ACH 100 or 200µg IC depending on the dose that previously provoked the coronary artery spasm (both microvascular and epicardial spasm).

SUMMARY:
The goal of this clinical trial is to assess the feasibility and clinical value of acetylcholine (ACH) rechallenge after intracoronary verapamil +- nitroglycerine in a patient cohort with angina and non-obstructive coronary arteries (ANOCA).

The main questions it aims to answer are:

* to determine the efficacy of these drugs in treating ACH-induced coronary artery spasm
* to determine the efficacy of these drugs in preventing ACH-induced coronary artery spasm

The ACH rechallenge will take place during the index coronary function tests in patients with proven ACH-induced vasospastic angina. The study is considered a feasibility study, no control arm is included.

ELIGIBILITY:
Inclusion Criteria:

* Clinically indicated coronary angiogram in the setting of angina with non-obstructive coronary artery disease (ANOCA)
* Non-obstructive coronary artery disease is defined as the absence of coronary artery stenosis ≥ 50%, or if ≥ 50% with non-ischemic resting (RFR > 0.89) and hyperemic indices (FFR > 0.80).
* ACH provoked epicardial and/or microvascular spasm
* Left ventricular ejection fraction (LVEF) > 50%
* Renal function with eGFR ≥ 40 ml/min

Exclusion Criteria:

* Obstructive coronary artery disease (both chronic and acute coronary coronary syndromes)
* Any cardiomyopathy (including takotsubo stress cardiomyopathy) or severe valvular disease
* LVEF < 50%
* Long QT syndrome (LQTS) - genetic or acquired
* Ventricular paced rhythm
* Renal failure with eGFR < 40 ml/min
* Thyroid stimulating hormone (TSH) < lower limit of normal (LLN). A subject taking thyroid replacement therapy may be enrolled with TSH level below LLN if, in the opinion of the investigator, the subject is in a clinically euthyroid state.
* Known hypersensitivity or contra-indication for either acetylcholine, verapamil, nicorandil or nitroglycerine.
* Pregnant female subjects. Female subjects of child-bearing potential should be on adequate contraceptive measures or are to be screened with a urine pregnancy test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01-09 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
The percent of ACH provoked spasm that is no longer inducible by ACH after IC injection of verapamil. | Baseline
  Is verapamil able to suppress ACH-induced coronary artery spasm?
The percent of ACH provoked spasm that is no longer inducible by ACH after sequential IC injection of verapamil and NTG. | Baseline
  Is verapamil + NTG able to suppress ACH-induced coronary artery spasm?

SECONDARY OUTCOMES:
The percent of ACH provoked spasm that resolves after IC administration of verapamil. | Baseline
  How efficient is verapamil IC as a treatment for ACH-induced coronary artery spasm?
The percent of ACH provoked spasm that resolves after sequential IC administration of verapamil and NTG. | Baseline
  How efficient is verapamil and NTG IC as a treatment for ACH-induced coronary artery spasm?

OTHER OUTCOMES:
Proportion of patients with epicardial coronary artery spasm who have microvascular spasm after either verapamil or verapamil + NTG. | Baseline
  Do microvascular and epicardial vasospasm occur simultaneously and is it possible to unmask microvascular spasm with either verapamil or verapamil + NTG.
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0 | Baseline
  Are there safety concerns related to the proposed ACH rechallenge protocol?
Absolute changes in the individual, overall and summary score of the Seattle Angina Questionnaire (SAQ) from baseline to the first ambulatory control visit. | Baseline, 1 month
  Does treatment based on the current protocol improve control of angina at the first ambulatory visit compared to before the coronary function tests?

CONTACTS AND LOCATIONS:
Overall Officials: Tijs Bringmans, Principal Investigator — University Hospital, Antwerp
Locations (1):
- University Hospital Antwerp, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No